CLINICAL TRIAL: NCT04873323
Title: A Study to Evaluate the Effects on QT/QTc Interval of TS-142 in Healthy Adult Subjects
Brief Title: A QT/QTc Evaluation Study of TS-142 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TS142-209
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — TS-142; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TS-142 10 mg (Experimental): TS-142 therapeutic dose oral tablet (low dose)
  Interventions: Drug: TS-142
- TS-142 30 mg (Experimental): Description: TS-142 supratherapeutic dose oral tablet (high dose)
  Interventions: Drug: TS-142
- Moxifloxacin 400 mg (Experimental): Moxifloxacin tablet
  Interventions: Drug: Moxifloxacin
- Placebo (Experimental): Placebo oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-142 — Single dose of TS-142 10 mg or TS-142 30 mg in the morning under fasting in each period
  Arms: TS-142 10 mg; TS-142 30 mg
Drug: Moxifloxacin — Single dose of moxifloxacin 400 mg in the morning under fasting in each period
  Arms: Moxifloxacin 400 mg
Drug: Placebo — Single dose of TS-142 placebo in the morning under fasting in each period
  Arms: Placebo

SUMMARY:
A clinical study to evaluate the effects on QT/QTc Interval of TS-142 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* Japanese Males or females aged 20 years or older but less than 40 years at the time of informed consent
* those with a BMI of 18.5 in male (17.6 in female) or more and less than 25.0 and a body weight of 40.0 kg or more at screening test
* those whose pulse rate measured by standard 12-lead ECG is 50 beats/min or more but no more than 90 beats/min at screening test and at the time before administration of investigational drug in period 1
* those who are judged eligible to participate in the study by the principal investigator or sub-investigator based on the results of screening test and test conducted before administration of investigational drug in period 1. However, if who showed abnormal findings but not clinically significant, they can be enrolled in clinical trials based on comprehensive consideration of medical viewpoints by the principal investigator or subinvestigator.
* those who are able to receive the explanation before participating in the study, understand the content of the study, and provide written informed consent by the subjects themselves.

Exclusion Criteria:

* Subjects who have any disease and are not considered healthy subjects based on the medical judgment of the principal investigator or sub-investigator.
* Subjects with a medical history considered inappropriate for participation in the study, including respiratory, cardiovascular, gastrointestinal, hepatic, renal, urological, endocrine, metabolic, hematological, immune, skin, neurological, and psychiatric diseases.
* Subjects with a history of drug allergy or food allergy.
* Subjects with a history of hypersensitivity to moxifloxacin or other quinolone antimicrobials
* Subjects with risk factors or with a history of risk factors for aortic aneurysm, aortic dissection (such as Marfan syndrome)
* Subjects with significant allergic predisposition (such as asthma requiring medical treatment)
* Subjects with congenital disease, heart disease, or a history of heart disease
* Subjects with risk factors or with a history of risk factors for torsade de pointes (TdP) (heart failure, hypokalemia, family history of long QT syndrome, etc.)
* Subjects with a history of unconscious seizures suspected of involving TdP.
* Subjects with waveforms difficult to assess for QTc interval prolongation in standard 12-lead ECG at screening and the timing before administration of investigational product in period 1 (drift, electromyography contamination, T-wave geometry, marked sinus arrhythmia, frequent premature beats, etc.)
* Subjects with QTcF(Fridericia correction method) of at least 450 msec in men and at least 470 msec in women in standard-12-lead ECG at screening test and at the time before administration of investigational product in period 1.
* Subjects with suicidal ideation, suicide attempt on the Colombian Suicide Assessment Scale (C-SSRS) on Day-1 or a history of suicide attempt within the previous 5 years.
* Other protocol defined inclusion criteria could apply

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
QTcF:QT-interval corrected by Fridericia corrections in Holter ECGs | Up to 24 hours postdose during each period
  Difference (ΔΔQTc) in change from baseline (ΔQTc) in QTc interval at each time point in each group compared with the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Direcoter, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Toshima-ku, Japan

IPD SHARING:
Plan to Share IPD: No